CLINICAL TRIAL: NCT02792660
Title: Identification of Cerebrospinal Fluid With Injeq IQ-Needle During Paediatric Lumbar Puncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Injeq Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INJ-SPINE-02
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Pediatric Lumbar Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Injeq IQ-Needle (Experimental): Lumbar puncture is performed using Injeq IQ-Needle
  Interventions: Device: Injeq IQ-Needle

INTERVENTIONS:
Device: Injeq IQ-Needle — Injeq IQ-Needle is a spinal needle that has bioimpedance measurement capability. It consists of traditional needle cannulae and removable bioimpedance probe which enables the measurement of bioimpedance. The needle is connected to measurement device and tissue identifying algorithm. Bioimpedance is measured during the operation and the algorithm detects when the needle tip is in contact with cerebrospinal fluid.

SUMMARY:
This is clinical feasibility study on the device performance with paediatric patients. The main objective is to validate the performance of investigational device in distinguishing and identifying the cerebrospinal fluid (CSF) inside the subarachnoid space during a lumbar puncture on paediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* Children whose diagnosis or treatment plan requires lumbar puncture to acquire a CSF sample.
* Consent from the parents

Exclusion Criteria:

* Being a high risk patient (as determined by the investigator)
* Any contraindication to a common lumbar puncture apply also in the investigation

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
Number of true/false positive and true/false negative detections of cerebrospinal fluid marked in case report form | During lumbar puncture
  Measurement device indicates with a sound and visual feedback when needle reaches cerebrospinal fluid (CSF). Physician verifies the location by removing the needle stylet and testing whether CSF flows from the needle, similarly as in traditional process. Detection is true positive if CSF flows from the needle and false positive if not. Even if the device does not detect CSF, physician performs the CSF test when needed. Physician marks to the case report form whether the device provided detections during the lumbar puncture and were the detections true or false detections.

CONTACTS AND LOCATIONS:
Overall Officials: Vesa Eskola, PhD MD, Principal Investigator — Tampere University Hospital
Locations (2):
- Finland (2):
  - Tampere University Hospital, Tampere
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: No